CLINICAL TRIAL: NCT00249691
Title: Medication Development for Cocaine Dependence
Brief Title: Effectiveness of Topiramate in Treating Cocaine Dependent Individuals - 1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bankole Johnson (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Bankole Johnson, Chair of Psychiatry and Neurobehavioral Sciences, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11578; R01DA017296 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2012-03-08 (Estimated); Status verified 2012-03

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine addiction; cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Topiramate; Cognitive Behavioral Therapy; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental)
  Interventions: Drug: Topiramate + Cognitive Behavioral Therapy
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo + Cognitive Behavioral Therapy

INTERVENTIONS:
Drug: Topiramate + Cognitive Behavioral Therapy — Topiramate up to 300 mg per day
  Other Names: Topamax
  Arms: Topiramate
Drug: Placebo + Cognitive Behavioral Therapy — Placebo twice a day
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
Although a great amount of research has been conducted to resolve cocaine dependence, an effective treatment has yet to be discovered. Topiramate is a drug that was found to be useful in treating alcohol dependence. The purpose of this study is to determine the effectiveness of topiramate in treating cocaine dependent individuals.

DETAILED DESCRIPTION:
Despite considerable scientific effort in the last two decades to develop treatment for cocaine dependent individuals, no medication has proven to be effective for treating cocaine dependence. Cocaine's rewarding effects are primarily a result of altering nerve pathways involving dopamine, a naturally-occurring chemical in the brain. Past research has focused on developing medications that either block dopamine or inhibit its release. However, these medications have not proven effective in treating cocaine dependence. This study will evaluate a new strategy of treating cocaine dependence by altering dopamine's functional expression. Dopamine-associated expression may be mediated through inhibition of gamma-aminobutyric acid (GABA), another brain chemical. Topiramate is a GABA inhibitor that has proven effective in treating alcohol dependent individuals. The purpose of this study is to determine the efficacy of topiramate in treating cocaine dependent individuals.

Participants will be randomly assigned to receive either 300 mg per day of topiramate or placebo. In addition, participants will receive weekly cognitive behavioral therapy for 12 weeks. Follow-up visits will occur at 2 weeks and 1, 2, and 3 months following completion of treatment, and will include evaluations of cocaine use and psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* Current DSM-IV diagnosis of cocaine dependence
* Good physical health as determined by a complete physical examination, an EKG within normal limits, and laboratory screening tests within acceptable parameters
* Seeking treatment for cocaine dependence
* At least one positive urine drug screen for cocaine at screen or baseline prior to randomization
* If female, a negative pregnancy test prior to study entry
* Agrees to use an effective method of contraception for the duration of the study
* Reads and writes English
* Willing to participate in behavioral treatment for cocaine dependence

Exclusion Criteria:

* Current DSM-IV diagnosis of dependence on any psychoactive substance other than cocaine, alcohol, nicotine, caffeine, or marijuana
* Physiological dependence on alcohol and requires medical detoxification
* Neurological or psychiatric disorders
* Any Axis 1 disorder that warrants treatment or would preclude safe participation
* Organic brain disease
* Dementia
* Bulimia and/or anorexia nervosa
* Seizure disorders or epilepsy
* Any disorder which would require ongoing treatment or which would make study agent compliance difficult
* History of suicide attempts and/or current suicidal ideation, as determined by the SCID, within the 30 days prior to screening
* Serious medical illnesses
* Mandated by the court to obtain treatment for cocaine dependence
* Expected to relocate from the study area
* AIDS diagnosis
* HIV with a CD4 positive T cell count less than 500 mm
* Any subjects on any pharmacotherapy for the treatment of AIDS or HIV will be excluded
* Active syphilis that has not been treated, or refused treatment for syphilis
* Severe or life-threatening adverse reactions to medications (including topiramate) in the past or during this clinical trial
* Currently receiving active treatment with topiramate
* Use of a drug with known potential for toxicity to a major organ system (e.g., isoniazid, methotrexate), within 30 days prior to study entry
* Pregnant or breastfeeding
* Concurrent regular use of psychotropics, including but not limited to antidepressants, anxiolytics, antipsychotics, anticonvulsants, and psychomotor stimulant-type medications, St. John's Wort, yohimbine, ginko biloba, horehound, or any other central nervous system active herbal preparations
* Use of any opiate substitutes (e.g., methadone, levo-alpha acetyl methadol, buprenorphine), within the month prior to screening
* Clinically significant test results that, in the investigator's opinion, require immediate or urgent treatment
* Fever of unknown origin or neuroleptic malignant syndrome
* Serious medical co-morbidity requiring medical intervention or close supervision
* Received inpatient or outpatient treatment for cocaine dependence within the 4 weeks prior to study entry
* Past participation in a clinical trial utilizing topiramate
* Treatment with electroconvulsive therapy within the 3 months prior to study entry
* Member of the same household of an individual enrolled in the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2005-10; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of topiramate to reduce cocaine use(assessed by a combination of self-report of use and urine assays for benzoylecgonine, the major metabolite of cocaine). | Throughout the study (Visit 0 to Visit 12, and at 2 weeks, 1, 2, and 3 months following completion of treatment)

SECONDARY OUTCOMES:
Improved psychosocial functioning; measured throughout the study, and at 2 weeks and 1, 2, and 3 months following completion of treatment | measured throughout the study, and at 2 weeks and 1, 2, and 3 months following completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bankole Johnson, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - UVA CARE, Charlottesville, Virginia
  - UVA CARE Richmond, Richmond, Virginia

REFERENCES:
- [Derived] Khalifa NR, Gibbon S, Vollm BA, Cheung NH, McCarthy L. Pharmacological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007667. doi: 10.1002/14651858.CD007667.pub3. PMID 32880105
- [Derived] Johnson BA, Ait-Daoud N, Wang XQ, Penberthy JK, Javors MA, Seneviratne C, Liu L. Topiramate for the treatment of cocaine addiction: a randomized clinical trial. JAMA Psychiatry. 2013 Dec;70(12):1338-46. doi: 10.1001/jamapsychiatry.2013.2295. PMID 24132249